CLINICAL TRIAL: NCT01029600
Title: Arthroscopic Capsulotomy vs Arthrographic Distention With Steroid in the Treatment of Primary Frozen Shoulder. A Randomized Study
Brief Title: Surgery or Capsular Distention With Steroid in the Treatment of Primary Frozen Shoulder?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bergen Surgical Hospital (Other)
Collaborators: Haraldsplass Deaconess Hospital (Other); Haukeland University Hospital (Other)
Responsible Party: Dr. Ove Kr. Austgulen, Bergen Surgical Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/870
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Adhesive Capsulitis
Keywords: Randomized study capsulotomy vs distention with steroid
MeSH Terms: conditions — Bursitis | interventions — Joint Capsule Release; Dilatation; Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthroscopic Capsulotomy (Active Comparator): Arthroscopic capsular release
  Interventions: Procedure: Arthroscopic capsular release
- Distention with steroid (Active Comparator): Arthrographic distention with contrast, saline, steroid and local anaesthetic
  Interventions: Procedure: Distention with steroid

INTERVENTIONS:
Procedure: Arthroscopic capsular release — Surgical division of thickened capsule in the shoulder
  Arms: Arthroscopic Capsulotomy
Procedure: Distention with steroid — Intraarticular distention with steroid, saline, contrast and local anaesthetic
  Arms: Distention with steroid

SUMMARY:
The purpose of the study is to compare two different treatment regimens for primary frozen shoulder: Arthroscopic capsulotomy and arthrographic distention with steroid.

DETAILED DESCRIPTION:
Patients with primary frozen shoulder will be randomized to two different treatments and the outcome will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have understood all information about the project and must have signed the informed consent letter about participation in the study including rehabilitation and follow-up
2. The patients must have a history and clinical findings typical for primary frozen shoulder with globally reduced range of motion in the shoulder.

   * External rotation 20 degrees or less
   * Abduction 45 degrees or less
3. The patients must not be in phase 1 (inflammation phase)
4. Diabetics may be included
5. MRI must be taken to exclude other reasons for stiffness

Exclusion Criteria:

1. Other reasons for stiffness( cuff rupture, arthritis)
2. Posttraumatic or postoperative stiffness
3. Patients not suited for day surgery
4. Patients with a history of subacromial impingement before developing stiffness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-03 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Shoulder Function | 2 years

SECONDARY OUTCOMES:
Shoulder range of motion | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eirik J Solheim, MD, PhD, Study Chair — University of Bergen, Surgical Dept.; Leiv Hove, MD, PhD, Study Director — University of Bergen, Surgical Dept.
Locations (1):
- Haraldsplass Deaconess Hospital, Bergen, Hordaland, Norway

REFERENCES:
- [Background] Codman EA. The Shoulder: Rupture of the Supraspinatus Tendon and Other Lesions In or About the Subacromial Bursa. Boston: Thomas Todd Co; 1934.
- [Background] Bridgman JF. Periarthritis of the shoulder and diabetes mellitus. Ann Rheum Dis. 1972 Jan;31(1):69-71. doi: 10.1136/ard.31.1.69. No abstract available. PMID 5008469
- [Background] Moren-Hybbinette I, Moritz U, Schersten B. The clinical picture of the painful diabetic shoulder--natural history, social consequences and analysis of concomitant hand syndrome. Acta Med Scand. 1987;221(1):73-82. doi: 10.1111/j.0954-6820.1987.tb01247.x. PMID 2436441
- [Result] Grey RG. The natural history of "idiopathic" frozen shoulder. J Bone Joint Surg Am. 1978 Jun;60(4):564. No abstract available. PMID 670287
- [Result] Reeves B. The natural history of the frozen shoulder syndrome. Scand J Rheumatol. 1975;4(4):193-6. doi: 10.3109/03009747509165255. PMID 1198072
- [Result] Binder AI, Bulgen DY, Hazleman BL, Roberts S. Frozen shoulder: a long-term prospective study. Ann Rheum Dis. 1984 Jun;43(3):361-4. doi: 10.1136/ard.43.3.361. PMID 6742896
- [Result] Duplay ES. De la periarthrite scapulo-humérale et des raideurs de l'épaule qui en sont la conséquence. Arch Gen Med 1872;20:513-42.
- [Result] Dias R, Cutts S, Massoud S. Frozen shoulder. BMJ. 2005 Dec 17;331(7530):1453-6. doi: 10.1136/bmj.331.7530.1453. PMID 16356983
- [Result] Shaffer B, Tibone JE, Kerlan RK. Frozen shoulder. A long-term follow-up. J Bone Joint Surg Am. 1992 Jun;74(5):738-46. PMID 1624489
- [Result] Pal B, Anderson J, Dick WC, Griffiths ID. Limitation of joint mobility and shoulder capsulitis in insulin- and non-insulin-dependent diabetes mellitus. Br J Rheumatol. 1986 May;25(2):147-51. doi: 10.1093/rheumatology/25.2.147. PMID 3708230
- [Result] Bunker TD, Anthony PP. The pathology of frozen shoulder. A Dupuytren-like disease. J Bone Joint Surg Br. 1995 Sep;77(5):677-83. PMID 7559688